CLINICAL TRIAL: NCT03021538
Title: Randomized Clinical Trial of Intraoperative Extracorporeal Membrane Oxygenation (ECMO) Versus Cardiopulmonary Bypass (CPB) in Lung Transplantation
Brief Title: Bypass vs. Ecmo in Lung Transplantation (BELT)
Acronym: BELT
Status: Terminated | Type: Observational
Why Stopped: Failure to enroll
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Michael Zhen-Yu Tong, MD, Cardiac Surgeon, The Cleveland Clinic
Other Study IDs: 17-166
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Results first posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Lung Transplant; Complications
Keywords: Cardiopulmonary Bypass; Extracorporeal Membrane Oxygenation; Primary Graft Dysfunction; Hemorrhage; Mechanical Ventilator
MeSH Terms: conditions — Primary Graft Dysfunction; Hemorrhage | interventions — Extracorporeal Membrane Oxygenation; Cardiopulmonary Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cardiopulmonary Bypass: There will be 40 patients placed on cardiopulmonary bypass during lung transplantation.
  Interventions: Device: Cardiopulmonary Bypass
- Extracorporeal Membrane Oxygenation: There will be 40 patients placed on ECMO during lung transplantation.
  Interventions: Device: Extracorporeal Membrane Oxygenation

INTERVENTIONS:
Device: Extracorporeal Membrane Oxygenation — ECMO is used during lung transplant procedure
  Groups: Extracorporeal Membrane Oxygenation
Device: Cardiopulmonary Bypass — CPB is used during lung transplant procedure
  Groups: Cardiopulmonary Bypass

SUMMARY:
This study seeks to compare outcomes of 2 different methods of cardiopulmonary support during lung transplant surgeries.

DETAILED DESCRIPTION:
This study will compare use of extracorporeal membrane oxygenation (ECMO) and heart-lung bypass (CPB) during lung transplant procedures and their short and long term outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. The study population will be all patients requiring cardiopulmonary support while undergoing lung transplantation at our institution.

Exclusion Criteria:

1. Patients undergoing concomitant cardiac operations with indication for obligate use of cardiopulmonary bypass
2. Patient with specific anatomy that require full cardiac decompression such as severe pulmonary hypertension or large heart that are shifted severely into the left chest
3. Patients with high likelihood of significant pleural bleeding that will require returning the blood back into the cardiotomy reservoir
4. Patients bridged to transplant with ECMO
5. Cystic fibrosis/bronchiectasis/resistant infection patients where surgeon will need to remove both lungs prior to implantation
6. Patients who the surgeon feels would be better served with CPB rather than ECMO- These patients will be entered into a registry and followed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be all patients requiring cardiopulmonary support while undergoing lung transplantation at our institution.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tong, M.D., M.B.A., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoechter DJ, von Dossow V, Winter H, Muller HH, Meiser B, Neurohr C, Behr J, Guenther S, Hagl C, Schramm R. The Munich Lung Transplant Group: Intraoperative Extracorporeal Circulation in Lung Transplantation. Thorac Cardiovasc Surg. 2015 Dec;63(8):706-14. doi: 10.1055/s-0035-1556873. Epub 2015 Aug 20. PMID 26291747
- [Background] Ius F, Kuehn C, Tudorache I, Sommer W, Avsar M, Boethig D, Fuehner T, Gottlieb J, Hoeper M, Haverich A, Warnecke G. Lung transplantation on cardiopulmonary support: venoarterial extracorporeal membrane oxygenation outperformed cardiopulmonary bypass. J Thorac Cardiovasc Surg. 2012 Dec;144(6):1510-6. doi: 10.1016/j.jtcvs.2012.07.095. Epub 2012 Aug 31. PMID 22944092
- [Background] Bermudez CA, Shiose A, Esper SA, Shigemura N, D'Cunha J, Bhama JK, Richards TJ, Arlia P, Crespo MM, Pilewski JM. Outcomes of intraoperative venoarterial extracorporeal membrane oxygenation versus cardiopulmonary bypass during lung transplantation. Ann Thorac Surg. 2014 Dec;98(6):1936-42; discussion 1942-3. doi: 10.1016/j.athoracsur.2014.06.072. Epub 2014 Oct 22. PMID 25443002
- [Background] Machuca TN, Collaud S, Mercier O, Cheung M, Cunningham V, Kim SJ, Azad S, Singer L, Yasufuku K, de Perrot M, Pierre A, McRae K, Waddell TK, Keshavjee S, Cypel M. Outcomes of intraoperative extracorporeal membrane oxygenation versus cardiopulmonary bypass for lung transplantation. J Thorac Cardiovasc Surg. 2015 Apr;149(4):1152-7. doi: 10.1016/j.jtcvs.2014.11.039. Epub 2014 Nov 21. PMID 25583107

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cardiopulmonary Bypass | Extracorporeal Membrane Oxygenation
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cardiopulmonary Bypass: There will be 40 patients randomized to cardiopulmonary bypass during lung transplantation.
  Cardiopulmonary Bypass: CPB is used during lung transplant procedure
- Extracorporeal Membrane Oxygenation: There will be 40 patients randomized to ECMO during lung transplantation.
  Extracorporeal Membrane Oxygenation: ECMO is used during lung transplant procedure
- Total: Total of all reporting groups
Arm/Group | Cardiopulmonary Bypass | Extracorporeal Membrane Oxygenation | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 9
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (7) | 54 (9) | 60 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 2 | 2 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Need for Blood Transfusion
Description: Number of pRBC transfusion that resulted due to postoperative bleeding
Time Frame: 72 hours after surgery
Measure: Mean (Standard Deviation); unit: number of pRBC transfusions
Arm/Group | Cardiopulmonary Bypass | Extracorporeal Membrane Oxygenation
Number analyzed (Participants) | 6 | 7
number of pRBC transfusions | 4.8 (6.1) | 6 (6.2)

ADVERSE EVENTS:
Time Frame: Up to hospital discharge
Arm/Group | Cardiopulmonary Bypass | Extracorporeal Membrane Oxygenation
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 0/6 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/38/NCT03021538/Prot_SAP_000.pdf